CLINICAL TRIAL: NCT04153682
Title: Impact of a Strategy Combining the Rapid Polymerase Chain Reaction Platform FilmArray® and the Intervention of an Antimicrobial Stewardship Team in Hospital-acquired Pneumonia : a Randomized Controlled Trial.
Brief Title: Trial on a Strategy Combining Rapid Diagnostic Testing and Antimicrobial Stewardship to Improve Antibiotic Use in Patients With Hospital-acquired Pneumonia.
Acronym: SHARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180391
Record Dates: First submitted 2019-09-02; First posted 2019-11-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Hospital-acquired Pneumonia
Keywords: Antimicrobial stewardship; hospital-acquired pneumonia; syndromic approach; rapid diagnostic testing
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimicrobial stewardship (= AMS) (Active Comparator): Management of HAP according to current practice, including intervention of the AMS team.
  Interventions: Diagnostic Test: Antimicrobial stewardship
- Antimicrobial Stewardship + Rapid Diagnostic Testing (Experimental): Management of HAP including rapid diagnostic testing (FA-PP) and intervention of the AMS team.
  Interventions: Diagnostic Test: Rapid Diagnostic Testing; Diagnostic Test: Antimicrobial stewardship

INTERVENTIONS:
Diagnostic Test: Rapid Diagnostic Testing — Automated microbiological diagnostic device based on multiplex PCR analysis, allowing detection of multiple pathogens and resistance markers in one hour from invasive and non-invasive respiratory samples
  Other Names: Filmarray® Pneumonia Panel (FA-PP)
  Arms: Antimicrobial Stewardship + Rapid Diagnostic Testing
Diagnostic Test: Antimicrobial stewardship — After clinical examination, routine biological tests will be performed. This includes blood culture, direct examination and culture of invasive or noninvasive respiratory samples, urinary antigen tests for Legionella and Pneumococcus, Influenza PCR on nasopharyngeal swabs (during the influenza season).
  Other Names: AMS

SUMMARY:
Hospital-Acquired Pneumonia (HAP) is the second most frequent hospital-acquired infection in the US and Europe and accounts for a large proportion of antibiotics prescribed in hospitals. Conventional methods to identify causative microorganisms (virus, bacteria) are time-consuming and sometimes inaccurate, leading to inadequate treatment in a large proportion of HAP patients.

The FILMARRAY® Pneumonia Panel (FA-PP, bioMérieux) is an automated diagnostic device, allowing detection of multiple pathogens and resistance markers in one hour. Strategies combining rapid diagnostic testing and intervention of specialists in infectious diseases (i.e. antimicrobial stewardship -AMS - experts) showed significant synergistic impact on antibiotic use, mortality and costs in bloodstream infections.

The trial hypothesis is that a strategy combining antimicrobial stewardship and FA-PP improves quality of care in HAP patients, as compared to antimicrobial stewardship alone.

The trial will include patients hospitalized for ≥ 48 hours, aged 18 years or older, who have criteria of pneumonia: new lung infiltrate on a chest-x ray, plus evidence that the infiltrate is of an infectious origin (i.e. new onset of fever and/or purulent sputum and/or leukocytosis and/or decline in oxygenation).

After informed consent, participants will be randomly allocated to either the intervention or the control arm.

In the control arm, management of HAP patients will include clinical examination and conventional microbiological tests. Antibiotic choice will be discussed between AMS experts and the physician in charge of the patient.

In the intervention arm, in addition to the procedures above, the strategy will include rapid testing using the FA-PP on a respiratory specimen, obtained by either invasive or non-invasive sampling. No additional invasive procedures will be required for the study, and FA-PP will be performed on samples collected as part as routine care.

Investigators will visit the patient at inclusion, on day 3 and on day 30 (or at hospital discharge) to collect data on comorbidities, clinical outcomes, results of microbiological tests and antibiotics. At the end of follow-up, we will compare the number of days on broad-spectrum antibiotics, the incidence of negative outcomes, the length of stay and costs in the two arms.

The use of the FA-PP is expected to prompt early adjustment of antibiotic therapy, improve outcomes, decrease length of stay, and to reduce the use of broad-spectrum antibiotics. The antibiotic saving may reduce the selection pressure, incidence of colonization with multidrug-resistant bacteria and incidence of hospital-acquired superinfections, both at an individual and hospital level. Moreover, this trial relies on the intervention of multidisciplinary AMS teams that are currently being implemented in many health facilities. Their transversal position offers opportunities for recruitment of patients from a wide range of medical and surgical departments. This project evaluates the feasibility of clinical trials based on the intervention of these teams, and will provide a high level of evidence regarding their impact on the prognosis of patients, appropriate use of antibiotics, and antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Any patient hospitalized for ≥ 48 hours
* aged 18 years or older
* not mechanically-ventilated at time of onset of pneumonia symptoms
* Dated and signed inform consent - written informed consent of relative (trusted person, close family) in case of emergency procedure, by default emergency inclusion notified in medical file and pursuance consent sought
* Affiliation with a social security scheme

Criteria of pneumonia:

* New lung infiltrate on a chest-x ray plus
* Evidence that the infiltrate is of an infectious origin, i.e. new onset of fever (> 38.5°C) and/or purulent sputum and/or leukocytosis and/or decline in oxygenation

Exclusion Criteria:

* Patients with severe chronic bronchitis structural changes: very severe COPD (Global initiative for chronic Obstructive Lung Disease GOLD 4), cystic fibrosis
* Radiological evidence of thoracic empyema, pulmonary abcess
* Patient life expectancy < 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of days on broad-spectrum antibiotics at day 30 or end-of follow-up for 100 patients-days | Day 30 or hospital discharge (plus or minus 4 days)
  Number of days that a patient is on an antibiotic, regardless of dose. The list of broad-spectrum antibiotics was defined according to previous literature data.

SECONDARY OUTCOMES:
Overall antibiotic use | Day 30 or hospital discharge (plus or minus 4 days)
  Number of days on antibiotics per 100 patient-days
Duration of antibiotics for the HAP episode | up to 30 days
  Number of days on any antibiotic for the HAP episode
Mortality | up to 30 days
In-hospital length of stay | up to 24 weeks
  Number of days between admission and discharge
Incidence of Clostridium difficile colitis | Day 30 or hospital discharge (plus or minus 4 days)
  Number of patients with documented Clostridium difficile colitis per 100 patient-days.
  Clostridium difficile colitis is defined by clinical evidence of colitis (unexplained and new-onset ≥3 unformed stools) and positive microbiological test relying on the multistep algorithm routinely used in each investigating center and compliant with national and international standards.
Medical direct costs | Day 30 or hospital discharge (plus or minus 4 days)
  Costs of the FILMARRAY® Pneumonia panel (labor and consumables), Antibiotic costs, Total admission costs
Analytical performances of the FILMARRAY® Pneumonia panel compared to conventional methods | End of the study
  Number of discrepancies on Micro-organism identification and Antibiotic resistance

CONTACTS AND LOCATIONS:
Overall Officials: Solen Kernéis, MD, PhD, Principal Investigator — Antimicrobial Stewardship Team, Hôpitaux Universitaires Paris Centre, Université de Paris
Locations (8):
- France (8):
  - Hôpitaux Universitaires Henri Mondor, Créteil
  - CHRU Nancy, Nancy
  - Hôpitaux Universitaires Paris Centre (Cochin) - service Médecine Intensive - Réanimation, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hôpitaux Universitaires Paris Centre-Site Cochin, Paris
  - Hôpitaux Universitaires Paris Nord Val de Seine-Site Bichat (SMIT), Paris
  - Hôpitaux Universitaires Paris Nord Val de Seine - EPRI (Bichat), Paris
  - Hôpitaux Universitaires Paris Nord Val de Seine - MIR (Bichat), Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Messika J, Stoclin A, Bouvard E, Fulgencio JP, Ridel C, Muresan IP, Boffa JJ, Bachmeyer C, Denis M, Gounant V, Esteso A, Loi V, Verdet C, Prigent H, Parrot A, Fartoukh M. The Challenging Diagnosis of Non-Community-Acquired Pneumonia in Non-Mechanically Ventilated Subjects: Value of Microbiological Investigation. Respir Care. 2016 Feb;61(2):225-34. doi: 10.4187/respcare.04143. Epub 2015 Dec 8. PMID 26647452
- [Background] Gadsby NJ, Russell CD, McHugh MP, Mark H, Conway Morris A, Laurenson IF, Hill AT, Templeton KE. Comprehensive Molecular Testing for Respiratory Pathogens in Community-Acquired Pneumonia. Clin Infect Dis. 2016 Apr 1;62(7):817-823. doi: 10.1093/cid/civ1214. Epub 2016 Jan 7. PMID 26747825
- [Background] Davey P, Marwick CA, Scott CL, Charani E, McNeil K, Brown E, Gould IM, Ramsay CR, Michie S. Interventions to improve antibiotic prescribing practices for hospital inpatients. Cochrane Database Syst Rev. 2017 Feb 9;2(2):CD003543. doi: 10.1002/14651858.CD003543.pub4. PMID 28178770
- [Background] Bookstaver PB, Nimmich EB, Smith TJ 3rd, Justo JA, Kohn J, Hammer KL, Troficanto C, Albrecht HA, Al-Hasan MN. Cumulative Effect of an Antimicrobial Stewardship and Rapid Diagnostic Testing Bundle on Early Streamlining of Antimicrobial Therapy in Gram-Negative Bloodstream Infections. Antimicrob Agents Chemother. 2017 Aug 24;61(9):e00189-17. doi: 10.1128/AAC.00189-17. Print 2017 Sep. PMID 28630187
- [Derived] Kerneis S, Visseaux B, Armand-Lefevre L, Timsit JF. Molecular diagnostic methods for pneumonia: how can they be applied in practice? Curr Opin Infect Dis. 2021 Apr 1;34(2):118-125. doi: 10.1097/QCO.0000000000000713. PMID 33395094